CLINICAL TRIAL: NCT03476070
Title: Adolescent and Young Adult Cancer Patients: Cognitive Toxicity on Survivorship (ACTS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Associate Professor, National University of Singapore
Other Study IDs: CIRB Ref. No: 2017/3139
Record Dates: First submitted 2018-03-06; First posted 2018-03-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Lymphoma; Germ Cell Tumor; Cognitive Impairment
Keywords: Adolescents and Young Adults (AYA); breast cancer; lymphoma; germ cell tumor; cognitive impairment; survivorship; Singapore
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Neoplasms, Germ Cell and Embryonal; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood processed into plasma and buffy coat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AYA cancer patients: Patients (aged between 15-39) diagnosed with breast cancer, lymphoma or germ cell tumor
- Healthy controls: Healthy controls

SUMMARY:
This study aims to evaluate the prevalence, biological mechanism and survivorship impact of cognitive toxicity among adolescent and young adult (AYA) patients diagnosed with curable cancers. The hypothesis is that cognitive impairment is clinically significant among AYA cancer patients treated with chemotherapy and that there will be detectable structural and functional changes in the brain for this patient group.

DETAILED DESCRIPTION:
A prospective longitudinal cohort study will be conducted at National Cancer Centre Singapore (NCCS) and KK Women's and Children's Hospital (KKH) from April 2018 to April 2021. Eligible cancer patients aged between 15-39 years old will be recruited and followed up for a period of 12 months. In addition, healthy individuals will also be recruited into the control arm of the study. The prevalence of cognitive impairment will be assessed via objective cognitive functional assessments in the form of the Cambridge Neuropsychological Test Automated Battery (Cantab) test scores and Functional Assessement of Cancer-Therapy Cognitive Function (FACT-Cog v3.0). The overall cognitive performance and post-treatment health issues measured by the assessment tools used would be compared between AYA cancer patients and healthy controls at baseline and 6 months after baseline.

Other post-treatment health issues will be assessed in relation to cognitive impairment with a series of questionnaires including Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) for cancer-related fatigue, the Rotterdam Symptom Checklist (RSCL) for symptom burden, the Paediatrics Quality of Life Inventory (PedsQL 4.0) for psychosocial outcomes, InCharge questionnaire for perceived financial distress and a work/education questionnaire respectively.

To enhance the understanding of the biological mechanism behind cognitive impairment, levels of biomarkers and genetic determinants will also be correlated with overall cognitive impairment. Blood plasma samples drawn from patients will be assessed for Brain-derived neutrotrophic factor (BDNF) levels, hormone levels and pro-inflammatory cytokines such as IL-1β, IL-4, and IL-6 using multiplex immunoassay. MRI scans and relevant neuroimaging techniques will be used to assess structural changes and functional connectivities in brain. Lastly, wearable devices will be utilized to track activity and lifestyle data among AYA cancer patients to investigate on the extent of impact of cognitive impairment and to assess the feasibility of using these wearables devices to personalize symptom management.

Findings from this proposed study will enhance understanding of cognitive toxicity and post-treatment health issues faced by the AYA patient group, which will facilitate the development of effective interventions to better cope with their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* between 15-39 years of age
* newly diagnosed with breast cancer, lymphoma or germ cell tumor with treatment intent determined as curative by medical oncologist
* scheduled for chemotherapy with or without non-cranial radiotherapy
* no prior history of chemotherapy and/or radiotherapy
* able to read and understand English
* capable of giving informed consent (or obtaining parents' consent if required)

Exclusion Criteria:

* physically or mentally incapable of providing verbal/written consent
* diagnosed with primary or metastatic brain tumor(s) or relapsed disease
* treatment includes intrathecal or intraventricular chemotherapy
* evidence of psychosis or underlying neuropsychiatric illness that may impair cognitive abilities
* have immediate family member who is enrolled as in the healthy control arm
* any contraindication to MRI as stated in the study protocol including: pregnancy, metal fragments/implants in body, known claustrophobia, and non-removable metal orthodontic braces, metallic retainers and oral wires

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The proposed study will be a multicenter, prospective, longitudinal, observational study conducted at the National Cancer Centre Singapore (NCCS) and KK Women's and Children's Hospital (KKH).
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cognitive impairment in AYA cancer patients | 6 months post recruitment
  Compare the prevalence of overall cognitive impairment at 6 months from baseline, between AYA cancer patients and healthy controls. Cognitive impairment is measured by the overall cognitive performance using the objective computer-based Cambridge Neuropsychological Test Automated Battery (Cantab ®).

SECONDARY OUTCOMES:
Prevalence of impairment in each individual Cantab ® cognitive domain | 1 year post recruitment
  The objective computer-based Cambridge Neuropsychological Test Automated Battery (Cantab ®) measures the domains attention, memory, executive function, response speed and processing speed.
Prevalence of self-reported cognitive impairment | 1 year post recruitment
  Functional Assessment of Cancer Therapy-Cognition Function (FACT-Cog) a 37-item questionnaire which measures six cognitive domains: memory, concentration, mental acuity, verbal fluency, functional interference and multitasking ability. The response is based on the perceived cognitive function within the past 7 days using a 5-point Likert scale ranging from 0 as "never" to 4 as "several times a day". The individual subscales scores are summed to determine the FACT-Cog total score, ranging from 0 to 148, with higher scores indicating better cognitive functioning. Self-reported cognitive impairment is measured using the minimal clinically important difference of 10.6 points.
Incidence and trajectory of cancer-related fatigue | 1 year post recruitment
  Multi-dimensional Fatigue Symptom Inventory-Short Form (MSFI-SF) is a 30-item questionnaire to assess the five domains of fatigue: general, emotional, vigour, physical and mental. The total score of the questionnaire is obtained by subtracting vigor from the sum of all domains. It ranges from -24 to 96, with a higher total score indicating increased fatigue. Cancer-related fatigue is defined using the minimal clinically important difference of 10.8 points.
Extent of symptom burden | 1 year post recruitment
  Rotterdam Symptom Checklist (RSCL) is used to measure symptom-related distress. It It uses a 4-point Likert-type scales (not at all, a little, quite a bit, very much) and contains 39 items in four domains: physical symptom distress, psychological distress, activity level and overall global life quality. The higher the score, the higher the level of burden or impairment.
Psychosocial outcomes | 1 year post recruitment
  Pediatrics Quality of Life Inventory (PedsQL) will be used to measure health-related quality of life in adolescents, with domains to assess both physical and psychosocial health. The psychosocial health summary score ranges from 0-100, whereby a higher score suggests a better HRQOL.
Extent of Financial Distress | 1 year post recruitment
  The InCharge Financial Distress/Financial Well-Being Scale is an 8-item scale designed to assess perceived financial distress. The score is obtained by summing the number of points of each of the items and dividing the total by 8. The scale ranges from a continuum from 1 to 10 where 1 represents overwhelming financial distress/lowest financial well-being and 10 being no financial distress/highest financial well-being.
Biomarker levels in relation to cognitive impairment | 1 year post recruitment
  Patients' plasma samples will be assessed for levels of BDNF, hormones and cytokines (IL1b, IL4, IL6) using multiplex immunoassay kits.
Neuroimaging scans | 6 months post recruitment
  Neuroimaging using MRI (Functional-MRI, Diffusion Weighted, T1-Weighted and T2-Weighted sequences) will be used to determine functional and structural changes in brain such as gray matter volume, which are then correlated to cognitive impairment
Lifestyle and activity data | 1 year post recruitment
  Wearable devices will be used to track patients' lifestyle data such as steps per day, intensity and duration of exercise and caloric expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, Pharm D, Principal Investigator — National University of Singapore, National Cancer Centre Singapore
Locations (3):
- Singapore (3):
  - KK Women's and Children's Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - National University of Singapore, Singapore

REFERENCES:
- [Background] Sender L, Zabokrtsky KB. Adolescent and young adult patients with cancer: a milieu of unique features. Nat Rev Clin Oncol. 2015 Aug;12(8):465-80. doi: 10.1038/nrclinonc.2015.92. Epub 2015 May 26. PMID 26011488
- [Background] Nass SJ, Beaupin LK, Demark-Wahnefried W, Fasciano K, Ganz PA, Hayes-Lattin B, Hudson MM, Nevidjon B, Oeffinger KC, Rechis R, Richardson LC, Seibel NL, Smith AW. Identifying and addressing the needs of adolescents and young adults with cancer: summary of an Institute of Medicine workshop. Oncologist. 2015 Feb;20(2):186-95. doi: 10.1634/theoncologist.2014-0265. Epub 2015 Jan 7. PMID 25568146
- [Background] Tai E, Buchanan N, Townsend J, Fairley T, Moore A, Richardson LC. Health status of adolescent and young adult cancer survivors. Cancer. 2012 Oct 1;118(19):4884-91. doi: 10.1002/cncr.27445. Epub 2012 Jun 11. PMID 22688896
- [Background] Ahles TA, Root JC, Ryan EL. Cancer- and cancer treatment-associated cognitive change: an update on the state of the science. J Clin Oncol. 2012 Oct 20;30(30):3675-86. doi: 10.1200/JCO.2012.43.0116. Epub 2012 Sep 24. PMID 23008308
- [Background] Vardy J. Cognitive function in breast cancer survivors. Cancer Treat Res. 2009;151:387-419. doi: 10.1007/978-0-387-75115-3_24. No abstract available. PMID 19593525
- [Background] Cheung YT, Shwe M, Tan YP, Fan G, Ng R, Chan A. Cognitive changes in multiethnic Asian breast cancer patients: a focus group study. Ann Oncol. 2012 Oct;23(10):2547-2552. doi: 10.1093/annonc/mds029. Epub 2012 Mar 6. PMID 22396443
- [Background] Guy GP Jr, Yabroff KR, Ekwueme DU, Smith AW, Dowling EC, Rechis R, Nutt S, Richardson LC. Estimating the health and economic burden of cancer among those diagnosed as adolescents and young adults. Health Aff (Millwood). 2014 Jun;33(6):1024-31. doi: 10.1377/hlthaff.2013.1425. PMID 24889952
- [Background] Poort H, Kaal SEJ, Knoop H, Jansen R, Prins JB, Manten-Horst E, Servaes P, Husson O, van der Graaf WTA. Prevalence and impact of severe fatigue in adolescent and young adult cancer patients in comparison with population-based controls. Support Care Cancer. 2017 Sep;25(9):2911-2918. doi: 10.1007/s00520-017-3746-0. Epub 2017 May 20. PMID 28528350
- [Background] Zimmer P, Baumann FT, Oberste M, Wright P, Garthe A, Schenk A, Elter T, Galvao DA, Bloch W, Hubner ST, Wolf F. Effects of Exercise Interventions and Physical Activity Behavior on Cancer Related Cognitive Impairments: A Systematic Review. Biomed Res Int. 2016;2016:1820954. doi: 10.1155/2016/1820954. Epub 2016 Apr 10. PMID 27144158
- [Background] Treanor CJ, McMenamin UC, O'Neill RF, Cardwell CR, Clarke MJ, Cantwell M, Donnelly M. Non-pharmacological interventions for cognitive impairment due to systemic cancer treatment. Cochrane Database Syst Rev. 2016 Aug 16;2016(8):CD011325. doi: 10.1002/14651858.CD011325.pub2. PMID 27529826
- [Background] Cheung YT, Lim SR, Ho HK, Chan A. Cytokines as mediators of chemotherapy-associated cognitive changes: current evidence, limitations and directions for future research. PLoS One. 2013 Dec 5;8(12):e81234. doi: 10.1371/journal.pone.0081234. eCollection 2013. PMID 24339912
- [Background] Kronfol Z, Remick DG. Cytokines and the brain: implications for clinical psychiatry. Am J Psychiatry. 2000 May;157(5):683-94. doi: 10.1176/appi.ajp.157.5.683. PMID 10784457
- [Background] Wefel JS, Vardy J, Ahles T, Schagen SB. International Cognition and Cancer Task Force recommendations to harmonise studies of cognitive function in patients with cancer. Lancet Oncol. 2011 Jul;12(7):703-8. doi: 10.1016/S1470-2045(10)70294-1. Epub 2011 Feb 25. PMID 21354373
- [Background] Chan A, Yo TE, Wang XJ, Ng T, Chae JW, Yeo HL, Shwe M, Gan YX. Minimal Clinically Important Difference of the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) for Fatigue Worsening in Asian Breast Cancer Patients. J Pain Symptom Manage. 2018 Mar;55(3):992-997.e2. doi: 10.1016/j.jpainsymman.2017.10.014. Epub 2017 Oct 31. PMID 29097274
- [Derived] Trudeau J, Ng DQ, Sayer M, Tan CJ, Ke Y, Chan RJ, Chan A. Brain-derived neurotrophic factor and cytokines as predictors of cognitive impairment in adolescent and young adult cancer patients receiving chemotherapy: a longitudinal study. BMC Cancer. 2025 Jul 1;25(1):1045. doi: 10.1186/s12885-025-14430-3. PMID 40597835
- [Derived] Chan A, Cheng I, Wang C, Tan CJ, Toh YL, Ng DQ, Koh YQ, Zhou H, Foo KM, Chan RJ, Ho HK, Chew L, Farid M, Tannock I. Cognitive impairment in adolescent and young adult cancer patients: Pre-treatment findings of a longitudinal study. Cancer Med. 2023 Feb;12(4):4821-4831. doi: 10.1002/cam4.5295. Epub 2022 Oct 11. PMID 36221816